CLINICAL TRIAL: NCT03852069
Title: Impact of a Diet Rich in Inulin-type Fructans Combined With Inulin Supplementation on Gut Microbiota Composition and Metabolic Parameters in Obese Patients
Brief Title: Inulin-type Fructans-rich Vegetables, Obesity, Gut Microbiota
Acronym: Food4Gut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B403201422056
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 16 g maltodextrin/day + recipes based on vegetables poor in inulin-type fructans
  Interventions: Dietary Supplement: Placebo
- Inulin (Experimental): 16 g inulin/day + recipes based on vegetables rich in inulin-type fructans
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Patient receive inulin as dietary supplement (16g/d) in combination with dietary advice to restrict caloric intake and to enhance the consumption of inulin-rich vegetables
  Arms: Inulin
Dietary Supplement: Placebo — Patient receive maltodextrin as dietary supplement (16g/d) in combination with dietary advice to restrict caloric intake and to enhance the consumption of vegetables poor in inulin
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the effect of a diet based on ITF-rich vegetables in combination with purified ITF supplementation on weight management, metabolic alteration and gut microbiota composition. Obese patients were treated for 3 months and several parameters were measured before and after the study period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 30 kg/m²
* Caucasian
* Presence of at least one of the following comorbidity : prediabetes, diabetes, dyslipidemia, hypertension, steatosis.

Exclusion Criteria:

* Psychiatric problems or use of antipsychotic
* Consumption of antibiotics, pro/prebiotics, fibre dietary supplement, or any molecules that modifies the intestinal transit (<6 weeks)
* Pregnancy in progress or planified within 6 months
* Specific dietary practise (vegetarian, vegan,...)
* Specific dietary treatment (<6 weeks) (e.g. high protein diet)
* Type 1 diabetes
* Excessive alcohol consumption (>3 glasses/day)
* Inconclusive acceptability test (regarding the protocol of the intervention and the vegetables used in the protocol)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | Month 0 - Month 3
  Relative abundance (percent) of bacterial taxa will be assessed by 16S rRNA gene sequencing

SECONDARY OUTCOMES:
Anthropometry | Month 0 - Month 3
  height (cm)
Anthropometry | Month 0 - Month 3
  weight (kg)
Anthropometry | Month 0 - Month 3
  hip circumference and waist circumference (cm)
Anthropometry | Month 0 - Month 3
  Body mass index (BMI, kg/m2)
Anthropometry | Month 0 - Month 3
  Body composition by bioimpedance analysis (fat mass, fat free mass, kg)
Anthropometry | Month 0 - Month 3
  Body composition by CT scan analysis (fat and muscle areas, cm2)
Blood pressure | Month 0 - Month 3
  systolic and diastolic blood pressures (mm Hg)
Glucose homeostasis | Month 0 - Month 3
  glycemia (mg/dl) (fasted, after an oral glucose tolerance test)
Glucose homeostasis | Month 0 - Month 3
  insulinemia (mU/l) (fasted, after an oral glucose tolerance test)
Glucose homeostasis | Month 0 - Month 3
  C-peptide (pM)
Glucose homeostasis | Month 0 - Month 3
  glycated hemoglobin HbA1c (percent)
Glucose homeostasis | Month 0 - Month 3
  dipeptidyl-peptidase IV activity in the plasma (UI/l)
Lipid homeostasis | Month 0 - Month 3
  HLD-Cholesterol, triglycerides, total cholesterol, free fatty acids in the plasma (mg/dl)
Hepatic fibrosis and/or steatosis | Month 0 - Month 3
  hepatic enzymes in the plasma (AST, ALT, gamma-glutamyl transpeptidase, U/l)
Hepatic fibrosis and/or steatosis | Month 0 - Month 3
  Elasticity by Fibroscan (kPa)
Hepatic fibrosis and/or steatosis | Month 0 - Month 3
  controlled attenuation parameter (CAP) by Fibroscan (dB/m)
Eating behavior | Month 0 - Month 3
  Questionnaire for Eating Disorders Diagnosis (Q-EDD). The Q-EDD is a 50-items questionnaire based on Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV allowing the psychologist to diagnose eating disorders (anorexia nervosa, bulimia, binge eating), there is no quantitative result.
Eating behavior | Month 0 - Month 3
  Dutch Eating Behaviour Questionnaire (DEBQ).The DEBQ is a 33-items questionnaire assessing 3 distinct behaviour: emotional eating (13 items), external eating (10 items) and restrained eating (10 items). Each item is rated on a 5-point scale. A high score is observed when individual tended to eat more when submitted to emotional and external stimuli (for emotional and external eating subscales) or when he displayed elevated cognitive control on its eating behaviour (for the restrained eating subscale).
Mood and emotional competence | Month 0 - Month 3
  Positive and Negative Affect Schedule (PANAS, two subscale - positive and negative - from 10 to 50, higher score associated with higher positive and negative emotion respectively)
Mood and emotional competence | Month 0 - Month 3
  Scale of Positive and Negative Experience (SPANE, two subscale - positive and negative - from 6 to 30, higher score associated with higher positive and negative emotion respectively)
Mood and emotional competence | Month 0 - Month 3
  Profile of Emotional Competence (PEC, from 0 to 5, higher score associated with better emotional competence).
Cognition | Month 0 - Month 3
  computer-based tests of the flexibility, the working memory and the inhibition of participants. The measurements will be the time to complete the task on the computer as well as the number of errors.
Dietary intake | Month 0 - Month 3
  one-week recall questionnaire to evaluate the dietary intake (macronutrients, caloric intake)
Biomarkers of systemic inflammation | Month 0 - Month 3
  Cytokines levels (Il-1β; IL-8; IL-12p70; IL-17a; MCP1; TNFα; IFNγ) by multiplex immunoassay (all in pg/ml)
Gut peptides | Month 0 - Month 3
  Gut peptide (GLP-1, GIP, ghrelin, PP, leptin) multiplex immunoassay (all in pg/ml)
Metabolomics | Month 0 - Month 3
  metabolomic analysis of biological samples (urine, blood and/or stool)
Physical activity | Month 0 - Month 3
  IPAQ questionnaire (The IPAQ long form asks details about the specific types of activities undertaken within the four main domains (leisure time PA, domestic and gardening (yard) activities, work-related PA and transport-related PA). Computation of the total scores for the long form requires summation of the duration (in minutes) and frequency (days) for all the types of activities in all domains. Results allowed us to classify different levels of PA proposed by the questionnaire (total, low-moderate or high-intensity physical activities)

OTHER OUTCOMES:
Fecal microbial-derived metabolites | Month 0 - Month 3
  Long and short chain fatty acid and bile acid profiles (ng/mg feces or percent) considered as exploratory analyses not initially scheduled in the study but performed in the context of the FiberTAG project. Before inclusion of the study, all participants provided written informed consent stipulating that any research outside the context performed in the future could only be conducted after approval by an ethics committee. We obtained agreement from the ethical committee of Saint-Luc for those exploratory analyses
Biomarkers of gut integrity and inflammation | Month 0 - Month 3
  Fecal zonulin (ng/mg feces) considered as exploratory analyses not initially scheduled in the study but performed in the context of the FiberTAG project. Before inclusion of the study, all participants provided written informed consent stipulating that any research outside the context performed in the future could only be conducted after approval by an ethics committee. We obtained agreement from the ethical committee of Saint-Luc for those exploratory analyses
Biomarkers of gut integrity and inflammation | Month 0 - Month 3
  fecal albumin (ng/mg feces) considered as exploratory analyses not initially scheduled in the study but performed in the context of the FiberTAG project. Before inclusion of the study, all participants provided written informed consent stipulating that any research outside the context performed in the future could only be conducted after approval by an ethics committee. We obtained agreement from the ethical committee of Saint-Luc for those exploratory analyses
Biomarkers of gut integrity and inflammation | Month 0 - Month 3
  fecal calprotectin (ng/mg feces) considered as exploratory analyses not initially scheduled in the study but performed in the context of the FiberTAG project. Before inclusion of the study, all participants provided written informed consent stipulating that any research outside the context performed in the future could only be conducted after approval by an ethics committee. We obtained agreement from the ethical committee of Saint-Luc for those exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Thissen, Pr., Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hiel S, Gianfrancesco MA, Rodriguez J, Portheault D, Leyrolle Q, Bindels LB, Gomes da Silveira Cauduro C, Mulders MDGH, Zamariola G, Azzi AS, Kalala G, Pachikian BD, Amadieu C, Neyrinck AM, Loumaye A, Cani PD, Lanthier N, Trefois P, Klein O, Luminet O, Bindelle J, Paquot N, Cnop M, Thissen JP, Delzenne NM. Link between gut microbiota and health outcomes in inulin -treated obese patients: Lessons from the Food4Gut multicenter randomized placebo-controlled trial. Clin Nutr. 2020 Dec;39(12):3618-3628. doi: 10.1016/j.clnu.2020.04.005. Epub 2020 Apr 13. PMID 32340903
- [Result] Leyrolle Q, Cserjesi R, Mulders MDGH, Zamariola G, Hiel S, Gianfrancesco MA, Rodriguez J, Portheault D, Amadieu C, Leclercq S, Bindels LB, Neyrinck AM, Cani PD, Karkkainen O, Hanhineva K, Lanthier N, Trefois P, Paquot N, Cnop M, Thissen JP, Klein O, Luminet O, Delzenne NM. Specific gut microbial, biological, and psychiatric profiling related to binge eating disorders: A cross-sectional study in obese patients. Clin Nutr. 2021 Apr;40(4):2035-2044. doi: 10.1016/j.clnu.2020.09.025. Epub 2020 Sep 28. PMID 33023763
- [Derived] Moens de Hase E, Neyrinck AM, Rodriguez J, Cnop M, Paquot N, Thissen JP, Xu Y, Beloqui A, Bindels LB, Delzenne NM, Van Hul M, Cani PD. Impact of metformin and Dysosmobacter welbionis on diet-induced obesity and diabetes: from clinical observation to preclinical intervention. Diabetologia. 2024 Feb;67(2):333-345. doi: 10.1007/s00125-023-06032-0. Epub 2023 Oct 28. PMID 37897566
- [Derived] Rodriguez J, Neyrinck AM, Van Kerckhoven M, Gianfrancesco MA, Renguet E, Bertrand L, Cani PD, Lanthier N, Cnop M, Paquot N, Thissen JP, Bindels LB, Delzenne NM. Physical activity enhances the improvement of body mass index and metabolism by inulin: a multicenter randomized placebo-controlled trial performed in obese individuals. BMC Med. 2022 Mar 30;20(1):110. doi: 10.1186/s12916-022-02299-z. PMID 35351144
- [Derived] Leyrolle Q, Cserjesi R, Demeure R, Neyrinck AM, Amadieu C, Rodriguez J, Karkkainen O, Hanhineva K, Paquot N, Cnop M, Cani PD, Thissen JP, Bindels LB, Klein O, Luminet O, Delzenne NM. Microbiota and Metabolite Profiling as Markers of Mood Disorders: A Cross-Sectional Study in Obese Patients. Nutrients. 2021 Dec 29;14(1):147. doi: 10.3390/nu14010147. PMID 35011021
- [Derived] Nachit M, Lanthier N, Rodriguez J, Neyrinck AM, Cani PD, Bindels LB, Hiel S, Pachikian BD, Trefois P, Thissen JP, Delzenne NM. A dynamic association between myosteatosis and liver stiffness: Results from a prospective interventional study in obese patients. JHEP Rep. 2021 Jun 15;3(4):100323. doi: 10.1016/j.jhepr.2021.100323. eCollection 2021 Aug. PMID 34355155
- [Derived] Neyrinck AM, Rodriguez J, Zhang Z, Seethaler B, Sanchez CR, Roumain M, Hiel S, Bindels LB, Cani PD, Paquot N, Cnop M, Nazare JA, Laville M, Muccioli GG, Bischoff SC, Walter J, Thissen JP, Delzenne NM. Prebiotic dietary fibre intervention improves fecal markers related to inflammation in obese patients: results from the Food4Gut randomized placebo-controlled trial. Eur J Nutr. 2021 Sep;60(6):3159-3170. doi: 10.1007/s00394-021-02484-5. Epub 2021 Feb 5. PMID 33544206
- [Derived] Leyrolle Q, Cserjesi R, D G H Mulders M, Zamariola G, Hiel S, Gianfrancesco MA, Portheault D, Amadieu C, Bindels LB, Leclercq S, Rodriguez J, Neyrinck AM, Cani PD, Lanthier N, Trefois P, Bindelle J, Paquot N, Cnop M, Thissen JP, Klein O, Luminet O, Delzenne NM. Prebiotic effect on mood in obese patients is determined by the initial gut microbiota composition: A randomized, controlled trial. Brain Behav Immun. 2021 May;94:289-298. doi: 10.1016/j.bbi.2021.01.014. Epub 2021 Jan 28. PMID 33515740